CLINICAL TRIAL: NCT00707590
Title: Randomized, Double-Blind, Placebo-Controlled Ascending Single and Multiple Dose Study to Evaluate the Safety, Tolerability, Pharmacokinetics, and Pharmacodynamics of BMS-767778 in Healthy Subjects and Subjects With Type 2 Diabetes Mellitus
Brief Title: Safety Study to Evaluate BMS-767778 in Healthy Subjects and Subjects With Type 2 Diabetes Mellitus (T2DM)
Status: Terminated | Phase: Phase 1 | Type: Interventional
Sponsor: Bristol-Myers Squibb (Industry)
Responsible Party: Study Director, Bristol-Myers Squibb
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: MB116-001
Record Dates: First submitted 2008-06-27; First posted 2008-07-01 (Estimated); Last update posted 2009-02-10 (Estimated); Status verified 2009-02

CONDITIONS: Type 2 Diabetes Mellitus
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — 2-(3-(aminomethyl)-4-(2,4-dichlorophenyl)-2-methyl-5-oxo-5H-pyrrolo(3,4-b)pyridin-6(7H)-yl)-N,N-dimethylacetamide

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- Part A (Experimental): A: BMS-767778, Oral Solution, Oral, 1 mg, once daily, 1 day OR Placebo Comparator, Oral Solution, Oral, 0 mg, once daily, 1 day
  B: BMS-767778, Oral Solution, Oral, 3 mg, once daily, 1 day OR Placebo Comparator, Oral Solution, Oral, 0 mg, once daily, 1 day
  C: BMS-767778, Capsules, Oral, 10 mg, once daily, 1 day OR Placebo Comparator, Capsules, Oral, 0 mg, once daily, 1 day
  D: BMS-767778, Capsules, Oral, 30 mg, once daily, 1 day OR Placebo Comparator, Capsules, Oral, 0 mg, once daily, 1 day
  E: BMS-767778, Capsules, Oral, 100 mg, once daily, 1 day OR Placebo Comparator, Capsules, Oral, 0 mg, once daily, 1 day
  F: BMS-767778, Capsules, Oral, 300 mg, once daily, 2 days OR Placebo Comparator, Capsules, Oral, 0 mg, once daily, 2 days
  G: BMS-767778, Capsules, Oral, 600 mg, once daily, 1 day OR Placebo Comparator, Capsules, Oral, 0 mg, once daily, 1 day
  Interventions: Drug: BMS-767778 or Placebo
- Part B (Experimental): A: BMS-767778, Capsules, Oral, 10 mg, once daily, 14 days OR Placebo Comparator, Capsules, Oral, 0 mg, once daily, 14 days
  B: BMS-767778, Capsules, Oral, 30 mg, once daily, 14 days OR Placebo Comparator, Capsules, Oral, 0 mg, once daily, 14 days
  C: BMS-767778, Capsules, Oral, 100 mg, once daily, 14 days OR Placebo Comparator, Capsules, Oral, 0 mg, once daily, 14 days
  D: BMS-767778, Capsules, Oral, 300 mg, once daily, 14 days OR Placebo Comparator, Capsules, Oral, 0 mg, once daily, 14 days
  E: BMS-767778, Capsules, Oral, 600 mg, once daily, 14 days OR Placebo Comparator, Capsules, Oral, 0 mg, once daily, 14 days
  Interventions: Drug: BMS-767778 or Placebo
- Part C (Experimental): A: BMS-767778, Capsules, Oral, Adaptive design (between 10 to 600 mg), 14 days OR Placebo Comparator, Capsules, Oral, 0 mg, 14 days
  B: BMS-767778, Capsules, Oral, Adaptive design (between 10 to 600 mg), 14 days OR Placebo Comparator, Capsules, Oral, 0 mg, 14 days
  Interventions: Drug: BMS-767778 or Placebo

INTERVENTIONS:
Drug: BMS-767778 or Placebo

SUMMARY:
To assess the safety and tolerability and the PK/PD relationship of BMS-767778 administered as single and multiple oral doses in healthy subjects, and in subjects with T2DM

ELIGIBILITY:
Parts A and Part B of the study (maximum age 45 years):

Inclusion Criteria:

* Healthy male and female subjects as determined by medical history, physical examination, 12-lead electrocardiogram (ECG), and clinical laboratory evaluations will be eligible to participate in the study.
* Men and women who are not of childbearing potential (i.e., who are postmenopausal or surgically sterile)

Exclusion Criteria:

* Evidence of organ dysfunction or any clinically significant deviation from normal in physical examination, vital signs, ECG or clinical laboratory determinations

Part C of the study (maximum age 65 years):

Inclusion criteria:

* Drug naive patients with T2DM or patients who are on metformin-monotherapy (at current dose for ≥ 8 weeks) with inadequately controlled blood glucose levels (HbA1c >7 %and <10 %) Men and women who are not of childbearing potential (i.e., who are postmenopausal or surgically sterile)

Exclusion criteria:

* Poorly controlled diabetes with either new onset or worsening of symptoms of polyuria and polydipsia, weight loss, fatigue, abdominal pain, or other significant signs and symptoms
* Any of the following medical conditions: uncontrolled hypertension, unstable angina pectora, Cushing's syndrome, Addison's disease, uncontrolled hyperthyroidism or hypothyroidism, significant liver disease or renal failure, malignant diseases, or immunodeficiency (e.g., HIV/AIDS or organ-transplant), or history of myocardial infarction, congestive heart failure defined as New York Heart Association (NYHA) stage II and above, significant valvular disease, cardiac arrhythmia, or transient ischemic attack or cerebrovascular accidents (occurred within 6 months prior to entry into the study), or family history of Long QT Syndrome

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2008-08; Primary Completion 2008-11 (Actual); Study Completion 2008-11 (Actual)

PRIMARY OUTCOMES:
AEs, vital signs, ECG and clinical laboratory test results | throughout the study

SECONDARY OUTCOMES:
Single and multiple dose (14 days) PK | throughout the study
DPP-4 inhibition and incretin response | throughout the study

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (1):
- Local Institution, Québec, Quebec, Canada